CLINICAL TRIAL: NCT04951323
Title: Impact of the Immune System on Response to COVID-19 Vaccine in Allogeneic Stem Cell Recipients (Covid Vaccin Allo)
Brief Title: Impact of the Immune System on Response to Anti-Coronavirus Disease 19 (COVID-19) Vaccine in Allogeneic Stem Cell Recipients (Covid Vaccin Allo)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Frédéric Baron, Professor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TJB2101
Record Dates: First submitted 2021-06-02; First posted 2021-07-06 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Coronavirus Disease 2019 (Covid19); Hematopoietic Neoplasms
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms | interventions — BNT162 Vaccine; CVnCoV COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection of anti-COVID19 mRNA-based vaccine (BNT162b2, Comirnaty®, commercialized by Pfizer) (Experimental): Injection of two doses (at Day 1 and Day 21) of the anti-COVID19 mRNA-based vaccine (BNT162b2, Comirnaty®, commercialized by Pfizer)
  Interventions: Drug: anti-COVID19 mRNA-based vaccine (BNT162b2, Comirnaty®, commercialized by Pfizer)

INTERVENTIONS:
Drug: anti-COVID19 mRNA-based vaccine (BNT162b2, Comirnaty®, commercialized by Pfizer) — Participants will receive the COVID-19 mRNA Vaccine BNT162b2 (Comirnaty®). The vaccine is administered intramuscularly after dilution as a series of two doses at least 21 days apart.
  Other Names: COVID-19 mRNA Vaccine; Pfizer

SUMMARY:
The present study is a prospective phase IV study. All participants will receive the anti-Coronavirus Disease 2019 (COVID-19) Vaccine (messenger Ribonucleic acid-based vaccine, BNT162b2 or Comirnaty®, commercialized by Pfizer-BioNTech) being authorized in the European Union since December 2020. The vaccine is administered intramuscularly after dilution as a series of two doses at least 21 days apart.

DETAILED DESCRIPTION:
The central question is whether allo-hematopoietic cell transplantation (allo-HCT) recipients can develop protective immunity against COVID-19 upon vaccination. This question needs to be answered urgently and would help the hematologist to provide recommendation / best treatment for these patients. In this pilot project Cov-Allo, this important question will be addressed in a cohort in which allo-HCT recipients will be vaccinated with the mRNA available COVID-19 vaccine according to the Belgian vaccination program. The primary objective is to assess immune response after administration of COVID-19 mRNA Vaccine BNT162b2 (Comirnaty®; Pfizer-BioNTech) in a population of 50 patients allo-HCT recipients. This number is based on the availabilities of vaccines and eligible patients. Moreover, as the study is observational and exploratory, no sample size calculation could be provided for this study.

ELIGIBILITY:
Inclusion Criteria:

* prior allogeneic hematopoietic stem cell transplantation 3 months to 5 years earlier (any donor type)
* age > or = 18 years at inclusion.
* written informed consent

Exclusion Criteria:

* HIV seropositivity
* Pregnancy
* Active malignant disease at inclusion
* Current grade III-IV acute Graft Versus Host Disease (GVHD)
* In vitro T-cell depletion of the graft if vaccination within the 6 months after transplantation.
* Rituximab administration in the 6 months prior to study inclusion
* Prior documented COVID-19 infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of anti-SARS-CoV-2 receptor binding domain specific IgG | Day 49 after first injection (D0)
  The primary endpoint is the quantification of different anti-SARS-CoV-2 specific IgG antibodies after vaccination (at Day 49) in allo-HCT recipients.

SECONDARY OUTCOMES:
Evolution of anti-SARS-CoV-2 receptor binding domain specific IgG | 6 months after day 21
  To study the evolution anti-RBD IgG titers from day +49 (day 28 after the second dose) to 6 months after the second dose.
Titration of neutralizing antibodies | Day 49 and 6 months after Day 21
  To analyze the titer of neutralizing antibodies at Day 49 as well as at 6 months after the second dose (at Day 21).
Clinical factors predicting response to vaccine (defined as detectable specific anti-SARS-CoV-2 RBD specific IgG). | 49 days after the first dose
  This point aims at trying to find correlations between patient immunity at vaccination and response to vaccination and also to correlate pre-vaccination clinical factors (such as delay from transplantation to vaccination in days, presence or not of moderate/severe chronic GVHD (assessed using the NIH criteria), administration of rituximab in the year before vaccination) response to the vaccine defined as detectable specific anti-SARS-CoV-2 RBD specific IgG.
Efficacy of the immune response to the vaccine to prevent COVID-19 | 12 months after first dose (Day 0)
  Incidence of SARS-CoV-2 infection occurring after vaccination
Assessment of T cell and B cell response to the vaccine | Day 7 and Day 49
  Measuring SARS-Cov2 specific T cells (by intracellular cytokine staining) and B cells (by Elispot).

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 12 months after first dose (Day 0)
  To investigate the safety of the anti-COVID-19 mRNA Vaccine (BNT162b2, Comirnaty®, Pfizer). Safety will be reported in terms of incidence and severity of systemic adverse events (AEs). Incidence and nature of newly occurring immune related Adverse Events of grade ≥ 3 according to the Common Terminology Criteria for Adverse Events version 5.0 including information on vaccine specific safety.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric MD Baron, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU Liège, Domaine du Sart-Tilman, Liège, Belgium